CLINICAL TRIAL: NCT01600963
Title: A Phase III Placebo-controlled, Double-blind, Randomized Trial to Evaluate the Efficacy and Safety of TMC207 in Subjects With Sputum Smear-positive Pulmonary Infection With Multi-drug Resistant Mycobacterium Tuberculosis (MDR-TB)
Brief Title: A Study to Evaluate the Efficacy and Safety of TMC207 in Patients With Pulmonary Infection With Multi-drug Resistant Mycobacterium Tuberculosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PhIII program revised; TMC207-C210 cancelled
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100807; TMC207-TIDP13-C210 (Other: Janssen Infectious Diseases BVBA); 2011-000653-23 (EudraCT Number); U1111-1135-7013 (Other: Universal Trial Number)
Record Dates: First submitted 2012-04-24; First posted 2012-05-17 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Multi-drug Resistant Tuberculosis
Keywords: Multi-drug resistant tuberculosis; Pre-extensively drug resistant tuberculosis; TMC207; Background regimen
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Arm A Double-blind Phase: TMC207; Drug: Treatment Failure During Double-blind Phase: TMC207; Drug: Treatment Failure During Follow-up Phase: TMC207
- Arm B (Placebo Comparator)
  Interventions: Drug: Arm B Double-blind Phase: Placebo; Drug: Treatment Failure During Double-blind Phase: TMC207; Drug: Treatment Failure During Follow-up Phase: TMC207

INTERVENTIONS:
Drug: Arm A Double-blind Phase: TMC207 — Type=exact number, unit=mg, number=400 mg for the first 2 weeks and 200 mg 3 times per week for the remainder of the treatment period, form=tablet, route=oral administration.
  Arms: Arm A
Drug: Arm B Double-blind Phase: Placebo — Form=tablet, route=oral administration, taken once daily for 2 weeks then 3 times per week for the remainder of the treatment period.
  Arms: Arm B
Drug: Treatment Failure During Double-blind Phase: TMC207 — Type=exact number, unit=mg, number=200 mg 3 times per week, form=tablet, route=oral administration.
Drug: Treatment Failure During Follow-up Phase: TMC207 — Type=exact number, unit=mg, number=400 mg once daily for 2 wks and 200mg three times per week for 22 weeks, form=tablet, route=oral administration.

SUMMARY:
The purpose of this study is to provide safety and efficacy data for TMC207 and to demonstrate that TMC207 added to a background regimen (BR) is superior to treatment with the BR plus placebo.

DETAILED DESCRIPTION:
This is a randomized (individuals will be assigned by chance to study treatments), double-blind (individual and investigator will not know the identity of study treatments), placebo (substance containing no active medication)-controlled, 2-arm study in patients with sputum smear-positive pulmonary infection with multi-drug resistant tuberculosis (MDR-TB) defined as tuberculosis (TB) due to infection with a strain of Mycobacterium tuberculosis (M. tuberculosis) that is resistant to both isoniazid and rifampin, or pre-extensively drug resistant (pre-XDR-TB) defined as TB due to infection with an MDR strain of M. tuberculosis that is resistant either to at least one of the injectable second-line drugs [amikacin, kanamycin, or capreomycin] or to any fluoroquinolone, but not both). Approximately 600 patients with sputum smear-positive pulmonary infection with MDR-TB or pre-XDR TB will receive a background regimen (BR) of MDR-TB therapy and will be randomly assigned in a 1:1 ratio to one of 2 treatment arms (Arms A [TMC207 + BR] and B [placebo + BR]). All patients will receive TMC207 or placebo in combination with a BR of MDR-TB therapy. TMC207 (or matching placebo) will be taken as oral tablets at a once daily dose of 400 mg for the first 2 weeks and 200 mg 3 times/week for the remaining period of TMC207 (or matching placebo) administration. The study will consist of a screening phase of a maximum of 3 weeks, a 36-week double-blind treatment phase, followed by a 48-week follow-up phase up to Week 84, also referred to as the treatment-free follow-up. After the treatment-free follow-up phase, there will be a safety follow-up phase of 48 weeks up to Week 132. Patients from Arms A or B who fail treatment according to prespecified criteria will be given the option to receive 24 weeks of TMC207 plus an individualized salvage regimen taken for a duration consistent with national TB guidelines. Efficacy and pharmacokinetic evaluations will be performed at time points as detailed in the protocol. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with sputum smear-positive pulmonary Mycobacterium multi-drug resistant tuberculosis; including pre-extensively drug resistant TB, and positive for acid fast bacilli on direct smear examination of expectorated or induced sputum specimen (>=1+ smear positive within the preceding 3 weeks) at screening and also on Day -1

Exclusion Criteria:

* Has known infection with extensively drug resistant tuberculosis isolate
* Has a clinically significant active medical condition such as, but not limited to, hepatic, pancreatic, renal, cardiovascular, gastrointestinal, hematologic, neurologic, locomotor, immunologic, ophthalmologic (e.g., corneal opacification or ulcers, uveitis, chorioretinitis), metabolic (except stable diabetes based on the investigator's judgement), endocrine, oncological disease, muscular disease (e.g., myositis, rhabdomyolysis), or psychiatric, dermatological illness, or any other illness that the investigator considers should exclude the patient or that could interfere with the interpretation of the study results. Eligibility of patients with poorly controlled diabetes as indicated by hemoglobin A1c higher than the normal range at screening should be based on the investigators judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with favorable treatment outcome at Week 60 | Week 60

SECONDARY OUTCOMES:
Number of patients with confirmed culture conversion at Week 84 | Week 84
Number of patients with confirmed culture conversion at Week 60 or at time of trial discontinuation | Up to Week 132
The number of patients with development of pre-extensively drug-resistant tuberculosis and extensively drug-resistant tuberculosis | Up to Week 132
Time to sputum culture conversion | Up to Week 132
Number of patients with negative culture and smear for tuberculosis | Up to Week 132
Time to positive signal in Mycobacteria Growth Indicator Tube (MGIT960) | Up to Week 132
Number of patients with confirmed culture conversion by lung cavity status | Up to Week 132
Number of patients with confirmed culture conversion by geographic region | Up to Week 132
Number of patients with confirmed culture conversion by human immunodeficiency virus status | Up to Week 132
Number of patients with confirmed culture conversion by baseline resistance to anti-tuberculosis therapy | Up to Week 132
Number of patients with Tuberculosis Symptom Profile symptoms at Week 36 and at the end of the treatment-free follow up | Up to Week 132
Number of tuberculosis-related deaths per investigator assessment | Up to Week 132
Number of patients with weight gain (greater than 5 percent) at Week 36 and at the end of the treatment-free follow up | Up to Week 132
Number of patients with improvements in laboratory assessments at Week 36 and at the end of the treatment-free follow up | Up to Week 132
Number of patients with improvements in chest radiograph assessments at Week 36 and at the end of the treatment-free follow up | Up to Week 132
Number of patients that received salvage regimen with favorable treatment outcome 24 weeks after the end of the individualized salvage regimen | Up to Week 132
Mean plasma concentrations of TMC207 | Up to Week 36
Mean plasma concentrations of N-monodesmethyl metabolite of TMC207 | Up to Week 36
Number of patients affected by an adverse event | Up to Week 132
Number of patients with confirmed culture conversion at Week 36 | Up to Week 132
Number of patients who required lung surgeries (resection or pneumonectomy) during the study | Week 84
Number of patients with confirmed culture conversion by baseline albumin grade | Up to Week 132
Number of patients with confirmed culture conversion by baseline TMC207 minimal inhibitory concentration | Up to Week 132
  Minimal inhibitory concentration is defined as lowest concentration of an antimicrobial agent that will inhibit the visible growth of an organism.
Number of patients with confirmed culture conversion at Week 132 | Week 132
Number of patients who required lung surgeries (resection or pneumonectomy) during the study | Week 132
Number of patients who experienced death | Up to Week 132
Number of patients will be qualified as cure based on the WHO outcome definition and the number of treatment failures, deaths, transfer out/defaults, and treatment completed | Up to Week 132
  Cure is defined as an multidrug-resistant tuberculosis (MDR-TB) patient who has completed the study procedures according to the protocol and has at least five consecutive negative cultures from samples collected at least 30 days apart in the final 12 months of the study. If only one positive culture is reported during that time, a patient may still be considered cured, provided that this positive culture is followed by a minimum of 3 consecutive negative cultures taken at least 30 days apart. Treatment failure is defined as a patient who completed the study procedures and was not cured as per the "Cure" definition based on the WHO classification during the study procedures. Defaults is defined as patients who discontinued study procedures for any reason. Treatment completed is defined as an MDR-TB patient who has completed the study procedures but does not meet the definition for cure or treatment failure due to lack of bacteriologic results.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (44):
- Brazil (3):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Phnom Penh, Cambodia
- China (7):
  - Beijing
  - Changsha
  - Chongqing
  - Fuzhou
  - Jinan
  - Nanjing
  - Shanghai
- Estonia (2):
  - Kohtla-Järve
  - Talinn
- Ethiopia (2):
  - Addis Ababa
  - Gonder
- Tbilisi, Georgia
- Stopinu Region, Latvia
- Monterrey, Mexico
- Lima, Peru
- Quezon City, Philippines
- Russia (6):
  - Arkhangelsk
  - Moscow
  - Novosibirsk
  - Oryol
  - Saint Petersburg
  - Yekaterinburg
- South Africa (3):
  - Paarl
  - Sandringham
  - Ysterplaat
- South Korea (6):
  - Busan
  - Daegu
  - Gwangju
  - Gyeongsangnam-Do
  - Incheon
  - Seoul
- Taiwan (4):
  - Changhua County
  - New Taipei City
  - Taichung
  - Tainan
- Nonthaburi, Thailand
- Keçiören, Turkey (Türkiye)
- Ukraine (3):
  - Donetsk
  - Kiev
  - Ternopil